CLINICAL TRIAL: NCT00428740
Title: Long-Term Intraocular Pressure Fluctuation and Visual Field Progression in Glaucoma Patients With Low Intraocular Pressure After Triple Procedure
Brief Title: Long-Term IOP Fluctuation and VF Progression After Triple Procedure
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Other Study IDs: 3-2006-0388
Record Dates: First submitted 2007-01-29; First posted 2007-01-30 (Estimated); Last update posted 2007-01-30 (Estimated); Status verified 2007-01

CONDITIONS: Glaucoma; Filtering Surgery; Intraocular Pressure
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Retrospective

SUMMARY:
Long-term intraocular pressure (IOP) fluctuation may be significantly associated with the progression of glaucomatous visual field loss, even in patients kept always low IOP after triple procedure, an effective approach for patients with coexisting glaucoma and visually significant cataracts.

DETAILED DESCRIPTION:
Previous studies reported that lowering intraocular pressure (IOP) slowed the advancement of visual field damage in glaucoma patients. However, even if the IOP can been substantially lowered, reduction of mean and peak IOP does not always prevent visual field progression.We believe that the long-term IOP fluctuation may play a significant role in visual field deterioration in those patients.

ELIGIBILITY:
Inclusion Criteria:

1. Underwent triple procedure
2. At leas 3 years of follow-up after surgery
3. IOP <18mmHg at each postoperative visit
4. A minimum of 5 visual field examinations
5. A reference visual field defect score of 16 or less
6. Good reliability indices of visual field

Exclusion Criteria:

1. Any other significant ocular diseases or intraocular surgical histories,
2. Diseases that may affect visual field or diabetes

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300
Dates: Start 2005-10; Study Completion 2005-12

CONTACTS AND LOCATIONS:
Overall Officials: Gong Je Seong, MD, PhD, Principal Investigator — Yondgong Severance Hospital, Yonsei University College of Medicine
Locations (1):
- Yonsei University College of Medicine, Seoul, South Korea

REFERENCES:
- [Derived] Hong S, Seong GJ, Hong YJ. Long-term intraocular pressure fluctuation and progressive visual field deterioration in patients with glaucoma and low intraocular pressures after a triple procedure. Arch Ophthalmol. 2007 Aug;125(8):1010-3. doi: 10.1001/archopht.125.8.1010. PMID 17698746